CLINICAL TRIAL: NCT03376139
Title: Zonisamide as a New Treatment for Post-Traumatic Stress Disorder and Co-Occurring Alcohol Use Disorder
Brief Title: Zonisamide Outpatient Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Pharmacotherapies for Alcohol and Substance Use Disorders Alliance (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS140026-A4; W81XWh-15-2-0077 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2017-11-13; First posted 2017-12-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Post Traumatic Stress Disorder; Alcohol Use Disorder
Keywords: Alcohol; Alcoholic; Alcoholism; Alcohol abuse; Alcohol Use Disorder; Alcohol use; Alcohol dependence; Alcohol dependent; PTSD; Post-Traumatic Stress Disorder; Veteran
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism; Alcohol Drinking | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted in a double-masked fashion in that both the participants and the site investigators and staff interacting with participants and assessing study outcomes will be masked to treatment assignment. The only individuals at the site with assess to treatment assignment information will be the research pharmacists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zonisamide (up to 400 mg/day) (Experimental): Zonisamide capsules titrated to a maximum tolerated dose of 400 mg/day for 35 days +/- 4 days, followed by a 14 day down-titration period.
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator): Encapsulated placebo filler (lactose) for 35 +/- 4 days, followed by a 14 day down-titration period. Placebo will go through a similar perceived titration process to maintain blind.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Zonisamide — Zonisamide capsules titrated to a maximum tolerated dose of 400 mg/day for 35 days +/- 4 days, followed by a 14 day down-titration period.
  Arms: Zonisamide (up to 400 mg/day)
Drug: Placebo Comparator — Encapsulated placebo filler (lactose) for 35 +/- 4 days, followed by a 14 day down-titration period. Placebo will go through a similar perceived titration process to maintain blind.
  Arms: Placebo

SUMMARY:
The objective of this study is to determine if, compared to placebo, zonisamide (400mg/day) is a safe and efficacious treatment for post-traumatic stress disorder (PTSD) and alcohol use disorder (AUD) in Veterans with PTSD and co-occurring AUD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to examine the ability of 5-weeks treatment with zonisamide to reduce symptoms of PTSD and AUD. The study population will consist of 60 Veterans with combat-related PTSD and co-morbid AUD. Veterans will be randomized 1:1 to receive either zonisamide (up to 400 mg/day) or placebo daily for 35±4days, followed by a 14-day down-titration period with follow-up. Primary efficacy variables are scores on the CAPS-5, fear-potentiated startle (FPS) responses, and percent of heavy drinking days (%HDD).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to sign and date an informed consent form
2. Be a military service member or Veteran
3. Male or female, 18-55 years of age
4. Meet Diagnostic and Statistical Manual (DSM)-5 criteria for AUD
5. Meet the DSM-5 diagnostic criteria for PTSD; PTSD diagnosis and severity will be determined based on CAPS-5 score greater than or equal to 33
6. Self-report drinking heavily (5 standard units for males, 4 for females) on at least 30% of the 42 days prior to the screening interview
7. Score less than 10 on the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar) assessed in the context of a breath alcohol concentration (BAC) less than or equal to 0.02% to demonstrate that they do not need medical detoxification (Sullivan et al. 1989)
8. Have blood lab tests assessed at screening with ranges falling within the acceptable limits as noted in the protocol.
9. Have normal vitals (heart rate 60-100 bpm, systolic blood pressure 90-140 mmHg and diastolic blood pressure 60-90 mmHg) and a baseline ECG that demonstrates clinically normal sinus rhythm, clinically normal conduction, normal QTc, and no clinically significant arrhythmias. Note that clinical judgement will be used when characterizing bradycardia among some healthy subject populations, for example, conditioned veterans. Thus, some individuals with bradycardia (i.e., heart rate less than 60 bpm) may be enrolled as determined by the admitting physician.
10. Have a self-reported medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician
11. Psychotropic medication free (with exception of SSRIs/SNRIs) for 7 or more days (or longer, depending on medication half-life) prior to enrollment
12. Be willing/able to stop use of any sleep medication for the duration of the study
13. Be willing to comply with all study procedures and be available for the duration of the study
14. Women must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or using double-mode form of contraception (i.e. barrier plus, e.g., birth control pills + intrauterine device, condoms + spermicide, etc.). Women can be receiving hormone replacement treatment (HRT) if the HRT dose has been stable for a period of at least 3 months
15. Women must provide negative urine pregnancy tests prior to randomization
16. Be willing to undergo a hearing test and be able to detect 500-2000 Hz tones at 40 dB or less.

Exclusion Criteria:

1. DSM-5 criteria for substance use disorders other than alcohol or nicotine or test positive for prescription or illegal drugs. Regarding marijuana/THC, an individual must test negative at the screening. If an individual's test is positive, they will be given a grace period where they will have the opportunity to return and test negative prior to being enrolled.
2. Be pregnant or nursing
3. Be taking blood pressure medications, psychotropics (with exception of SSRIs/SNRIs), drugs effecting the CNS, medications contraindicated with ethanol, any sulfonamide, or any other medication that could interact with study medications or alter the effects of alcohol.

   a. Note that participants may currently be seeking treatment (or already receiving a behavioral treatment) for AUD, but may not be taking medications used in the treatment of AUD (acamprosate, disulfiram, oral naltrexone, and extended-release injectable naltrexone, and topiramate)
4. Have neurological or psychiatric disorders other than PTSD or AUD (except mild/moderate depression succeeding PTSD). Examples include:

   1. Current psychosis, bipolar illness or major depression requiring treatment.
   2. Organic brain disease or dementia assessed clinical interview.
   3. History of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult.
   4. History of suicide attempts within the past year and/or current suicidal ideation/plan
5. Have evidence of untreated or unstable medical illness including: cardiovascular, neuroendocrine, autoimmune, renal, hepatic, or active HIV+, AIDS infection.
6. Have a history of medically adverse reactions to alcohol (e.g., loss of consciousness, chest pain, or epileptic seizure) or major alcohol-related medical complications requiring hospitalization (i.e. hepatitis or pancreatitis)
7. Have contraindication(s) to take the study medications such as renal or hepatic impairment, congenital metabolic disorders, or hypersensitivity/allergies to study drug or similar compounds
8. Have current epilepsy or evidence suggestive of seizure disorder
9. Have past brain injury/head trauma with current symptoms (e.g. not photophobic, dizziness, etc.) or past report of loss of consciousness (LOC) for greater than 30 minutes and/or have been blast-exposed or had LOC of greater than 1 minute and current post-concussive symptoms
10. Self-report more than thirty days abstinence from alcohol during the three months prior to enrollment/consent
11. Current signs of violence or aggression, assessed as part of the consent process
12. Participation in a pharmaceutical trial or exposure to any investigational drugs within 1 month of the screening visit
13. Hearing loss that would interfere with the FPS measures
14. Have any other illness, condition, or use medications (psychotropic or antiretroviral), which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total symptom severity score | Baseline to post-treatment (weeks 0, 3, 5, 7)
  CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. All symptoms are assessed on a five-point scale (0=Absent, 1=Mild/subthreshold, 2=Moderate/threshold, 3=Severe/markedly elevated, 4=Extreme/incapacitating). CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms, possible scores ranging from 0-80 with higher values indicating a worse symptom severity.
Percent change in fear-potentiated startle (FPS) responses from acquisition on day 1 to recall on day 35. | Baseline to post-treatment (weeks 1, 5, 7)
Change from baseline in the percent of heavy drinking days (%HDD) | Baseline to post-treatment (weeks 0-7)
  Timeline Follow-Back (TLFB) of self-report assessment of heavy drinking days over the course of the five-week study treatment.

SECONDARY OUTCOMES:
Severity and numbers of AEs | Baseline to post-treatment (weeks 0-7)
  All safety analyses will be performed using the safety population (i.e., as treated) unless otherwise specified. Rates, severity and relatedness of adverse events including serious adverse events, study drug-related adverse events, and deaths will be evaluated.
Treatment retention | Baseline to post-treatment (weeks 0-5)
  Retention will be assessed as a comparison count of participants at baseline and post-treatment.
Medication compliance | Baseline to post-treatment (weeks 0-5)
  We will use self-report and pill count. Overall percentage of pills taken will be calculated and reported.
Medication adherence | Baseline to post-treatment (weeks 0-5)
  To assess medication adherence, urine samples collected at study visits will be tested for riboflavin, using a quantitative assessment of fluorescence. Results will be summarized over time for the active treatment study group.
Blood pressure | Baseline to post-treatment (weeks 0-7)
  Systolic and diastolic blood pressure results will be summarized over the time of the study.
Heart rate | Baseline to post-treatment (weeks 0-7)
  Heart beats per minute will be summarized over the time of the study.
ECG abnormalities | Baseline to post-treatment (weeks 0-7)
  Frequency of ECG Summary results (i.e. Normal, Abnormal but clinically insignificant, or Abnormal and clinically significant) will be summarized over the time of the study.
Breath alcohol content (BAC) | Baseline to post-treatment (weeks 0-7)
  BAC as measured by an alcohol breathalyzer test, lower percentages indicating less alcohol breath content.
Subjective and psychometric effects of alcohol (e.g. mood, urge/craving) | Baseline to post-treatment (weeks 0-7)
  Alcohol Urge Questionnaire (AUQ) scores will be calculated, with higher scores reflecting higher craving.
Alcohol use measures | Baseline to post-treatment (weeks 1, 3, 7)
  Drinks per day including days abstained from drinking will be evaluated.
Presence and symptom assessments for PTSD | Baseline to post-treatment (weeks 0-7)
  PTSD Checklist for DSM-5 (PCL-5) scores will be calculated, with higher scores reflecting higher severity.
Change from baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) subscale scores: Criterion B (reexperiencing) | Baseline to post-treatment (Weeks 0, 3, 5, 7)
  CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. All symptoms are assessed on a five-point scale (0=Absent, 1=Mild/subthreshold, 2=Moderate/threshold, 3=Severe/markedly elevated, 4=Extreme/incapacitating). Criterion B is the sum of items 1-5 (scores range 0-20). A higher score indicates worse symptom severity.
Change from baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) subscale scores: Criterion C (Avoidance) | Baseline to post-treatment (Weeks 0, 3, 5, 7)
  CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. All symptoms are assessed on a five-point scale (0=Absent, 1=Mild/subthreshold, 2=Moderate/threshold, 3=Severe/markedly elevated, 4=Extreme/incapacitating). Criterion C is the sum of items 6 and 7 (scores range 0-8). A higher score indicates worse symptom severity.
Change from baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) subscale scores: Criterion D (negative alterations in cognitions and mood) | Baseline to post-treatment (Weeks 0, 3, 5, 7)
  CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. All symptoms are assessed on a five-point scale (0=Absent, 1=Mild/subthreshold, 2=Moderate/threshold, 3=Severe/markedly elevated, 4=Extreme/incapacitating). Criterion D is the sum of items 8-14 (scores range 0-28). A higher score indicates worse symptom severity.
Change from baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) subscale scores: Criterion E (hyperarousal) | Baseline to post-treatment (Weeks 0, 3, 5, 7)
  CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. All symptoms are assessed on a five-point scale (0=Absent, 1=Mild/subthreshold, 2=Moderate/threshold, 3=Severe/markedly elevated, 4=Extreme/incapacitating). Criterion E is the sum of items 15-20 (scores range 0-24). A higher score indicates worse symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
CDMRP has a policy to share and make available to the public the results and accomplishments of the activities that it funds. The PASA consortium plans to share de-identified data after final publication in a government-supported data repository.

REFERENCES:
- [Background] Acheson DT, Geyer MA, Baker DG, Nievergelt CM, Yurgil K, Risbrough VB; MRS-II Team. Conditioned fear and extinction learning performance and its association with psychiatric symptoms in active duty Marines. Psychoneuroendocrinology. 2015 Jan;51:495-505. doi: 10.1016/j.psyneuen.2014.09.030. Epub 2014 Oct 7. PMID 25444643
- [Background] Acheson DT, Feifel D, Kamenski M, Mckinney R, Risbrough VB. Intranasal oxytocin administration prior to exposure therapy for arachnophobia impedes treatment response. Depress Anxiety. 2015 Jun;32(6):400-7. doi: 10.1002/da.22362. Epub 2015 Mar 31. PMID 25826649
- [Background] Acheson D, Feifel D, de Wilde S, McKinney R, Lohr J, Risbrough V. The effect of intranasal oxytocin treatment on conditioned fear extinction and recall in a healthy human sample. Psychopharmacology (Berl). 2013 Sep;229(1):199-208. doi: 10.1007/s00213-013-3099-4. Epub 2013 May 5. PMID 23644911
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811